CLINICAL TRIAL: NCT06660849
Title: Predicting the Presence and Duration of Atrial Fibrillation From Cortical Lens Opacity
Brief Title: Atrial Fibrillation Duration and Cortical Lens Opacity
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Şahbender Koç, Associate Professor Cardiologist, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: AnkaraAtaturkSTRH
Record Dates: First submitted 2024-09-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation (AF); Cataract Cortical
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1 ,group 2: The patients' median age was 70 years. Patients with New York Heart Association class 1, 2, or 3 heart failure (HF) were included, regardless of the cause of HF. Both groups comprised patients with a similar number and duration of comorbidities that contributed to their CHA2DS2-VASc scores.

SUMMARY:
The prevalence of atrial fibrillation (AF) and the risk of stroke increase with a higher CHA2DS2-VASc score. Osmotic stress, which also contributes to cortical cataract formation, increases in the presence of diseases that raise the CHA2DS2-VASc score. Knowledge of AF duration is crucial because it heightens the risk of AF-related complications. This study investigated whether the presence of cortical cataracts, classified using the Lens Opacity Classification System (LOCS)stage, can predict the presence and duration of AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common type of heart rhythm disorder encountered in clinical settings and is associated with increased morbidity and mortality. The prevalence of AF and the risk of stroke increase with higher CHA2DS2-VASc scores . Cortical cataracts develop at the periphery of the lens and progress toward the center in a spoke-like pattern. The incidences of AF and cortical cataracts significantly increase with age .

Similar to subclinical AF, the initial onset of AF may go undetected, and the time required for AF to become permanent varies. Longer episodes of AF and higher CHA2DS2-VASc scores are strongly associated with an increased annual risk of stroke or systemic embolism , making it essential to estimate the duration of AF.

Cortical cataract stages can be easily identified and monitored through simple biomicroscopic examination. To our knowledge, no reliable method currently exists to predict the duration of AF of unknown onset. This study investigated the relationship between cortical cataract stages and the presence and duration of AF by analyzing p.osmolarity data and comparing it with the LAVI.

ELIGIBILITY:
Inclusion Criteria:

Atrial Fibrillation patients

Exclusion Criteria:

Advanced HF (New York Heart Association class 4), Decompensated HF Prior cataract surgery Diabetic ketoacidosis Alcohol use Severe hyponatremia [sodium level of < 125 mEq/L], Nephrotic syndrome Cirrhosis Hypothyroidism

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 400 patients: 200 patients without AF (100 female, 100 male) and 200 patients with AF (100 female, 100 male). The patients' median age was 70 years. Patients with New York Heart Association class 1, 2, or 3 heart failure (HF) were included, regardless of the cause of HF.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
cortical cataract opacification grading. | day1
  All participants underwent detailed eye examinations using a biomicroscope . Digital photographs of the lenses were then captured using a smartphone under retro-illumination. Due to its simplicity, the Lens Opacity Classification System 2 [LOCS 2-Cortical] was used to perform cortical cataract opacification grading.
LAVI (left atrial volume index)(ml/m2) | day1
  LAVI were measured using a GE Vivid N60 echocardiography system

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Sanatoryum TR Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Relationship between cortical cataract stages and the presence and duration of AF
Supporting Information: CSR
Time Frame: 1-2 mounts
Access Criteria: All data generated in this study are available upon request from the corresponding authors except patient lens photographs.